CLINICAL TRIAL: NCT03913052
Title: A Research on The Effects of Intra-articular Viscosupplement Application Containing Hyaluronic Acid, Chondroitin Sulfate and Glucosamine Compounds on the Isokinetic Muscle Test Values of Patients With 40-65 Years of Knee Osteoarthritis
Brief Title: Intra-articular Viscosupplement Application in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, TOMRIS DUYMAZ, Asst. Prof. Ph.D., Istanbul Bilgi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OA2018
Record Dates: First submitted 2019-04-08; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection (Experimental): Injection containing hyaluronic acid, chondroitin sulphate and glucosamine was performed once when the knee joint was in the supine position and the knee was in the extension.
  Interventions: Procedure: Intra-articular Viscosupplement Application

INTERVENTIONS:
Procedure: Intra-articular Viscosupplement Application — Injection containing hyaluronic acid, chondroitin sulphate and glucosamine is performed once when the knee joint was in the supine position and the knee is in the extension.
  Other Names: intra-articular injection

SUMMARY:
Knee osteoarthritis (OA) is one of the common diseases which causes pain and disability with increasing age. In developed countries, it is said to be one of the ten diseases which decreases functionality most.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is one of the common diseases which causes pain and disability with increasing age. In developed countries, it is said to be one of the ten diseases which decreases functionality most. With a prevalence between 22% - 39%, 7% of which are patients who are over 65 years old, and when examined world-wide, it is stated that knee OA is seen 18% of women and 9,6% of men. Knee OA is characterized by pain, and; functional loss and progressive mobility where motions are required a physical activity of lower extremity. The disease causes 80% of restriction of motions and 25% of restriction of daily life activities. Additionally, along with the loss of proprioception, it can be seen defects of static and dynamic postural stability and the loss of balance. The factors of disease cause reduced muscle strength, defects of functionality of muscles and reduced workout capacity. According to the radiographic classification of Kellgren and Lawrence, quadriceps muscle weakness is frequently seen without atrophy and pain in early phases of knee OA of which degree is 0 or 1. If the symptoms are accompanied by a knee pain, the weakness of muscles will show an increase more and cause dysfunction and progression of disease. An increase of force in the muscles of quadriceps and hamstring plays a positive role for stability and mobility of joints and pain tolerance.

In the literature, studies with intra-articular HA injection in the treatment of knee OA are frequently seen, but the number of studies about the co-injection of HA, CS and GA is scarcely any. At the same time, studies investigating the effect of intra-articular viscosupplementation injection on isokinetic muscle strength was not observed. Therefore, the investigators aimed at investigating the effects of HA, CS and GA injection on isokinetic quadriceps and hamstring muscle strengths in our study.

ELIGIBILITY:
Inclusion Criteria:

* being between 40-65 years of age,
* being diagnosed with Stage 3 and 4 knee OA according to the Kellgren-Lawrence classification

Exclusion Criteria:

* any lower extremity deformity (knee flexion contracture, knee hyperextension, varus and valgus deformities),
* septic arthritis, rheumatoid arthritis,
* major dysplasia,
* congenital anomalies, acromegaly, primary osteochondromatosis,
* Ehler-Danlos syndrome,
* neuropathic arthropathy,
* hyperparathyroidism, hypothyroidism,
* diabetes mellitus,
* active synovitis,
* severe knee traumas,
* previous surgery and in the last year,
* knee arthroscopy, injections and fracture history and pregnancy

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Biodex (System 3) isokinetic systems | 5 minutes
  Isokinetic test are measured with Biodex (System 3) for the measurement of quadriceps muscle strength before and 3 months after injection. Measurements are performed at angular speeds of 60°. Biodex (System 3) isokinetic systems are used to evaluate knee flexion angles and the muscle strengths applied at these angular velocities. The device is set to measure at angular speeds of 60°. Knee extension and flexion are requested and the best measurement is made. By this measurement, the effect of injection on quadriceps isokinetic muscle strength will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Tomri̇s Duymaz, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Tomri̇s Duymaz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No